CLINICAL TRIAL: NCT07179809
Title: Pilot Randomized Trial of a Virtual, Group-based Comprehensive Lifestyle Program for Women With Metastatic Breast Cancer: Exploring Dose of Support to Optimize Adherence
Brief Title: Group-based Comprehensive Lifestyle Program for Women With Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0951; NCI-2025-06338 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-08-31; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Demography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACLP Program (Experimental): Participants will take part in the ACLP alone
  Interventions: Other: Demographics/Lifestyle Survey
- ACLP Program + Learning Circles (Experimental): Participants will take part in the ACLP and Learning Circles
  Interventions: Other: Demographics/Lifestyle Survey
- ACLP Program + Learning Circles + Individual Health Coaching (Experimental): Participants will take part in the ACLP and in Learning Circles After participants complete the ACLP with Learning Circles, they will receive up to 6 individualized health coaching sessions.
  Interventions: Other: Demographics/Lifestyle Survey

INTERVENTIONS:
Other: Demographics/Lifestyle Survey — Participants will complete all sessions and instruments

SUMMARY:
The research study is to learn how the ACLP can best support patients with stable HR+/HER2- MBC.

DETAILED DESCRIPTION:
Primary Objective:

Assess the feasibility of delivering the ACLP, ACLP-LC, and ACLP-LC-IHC programs in stable HR+/HER2- MBC survivors. Feasibility criteria will include the percent of eligible patients who consent to participate (feasibility is defined as 30% of those approached and are eligible end up consenting) and study retention by the last follow-up (feasibility is defined as 50% of those randomized remaining in the study and who participated in at least 75% of online sessions). Our working hypothesis is that the provision of the evidence-based, mHeath ACLP with the Learning Circle support group, with or without individual health coaching, is feasible in patients with stable HR+/HER2- MBC.

Secondary Objectives:

1. Explore changes in targeted health behaviors of diet, exercise, and stress management.
2. Examine changes in patient-reported outcomes (PROs), including: QOL, fatigue, sleep disturbances, mental health, social support, mindfulness, and stages of change.
3. Examine if there are group differences in post-intervention albumin, vit D, and magnesium levels.

OUTLINE: Patients are first randomized to 1 of 3 groups.

GROUP 1 (ACLP): Patients receive an outline of tasks and complete ACLP interactive exercise and activity modules on their own over 8 weeks and receive calls weekly for 8 weeks.

GROUP 2 (ACLP-LC): Patients complete ACLP interactive exercise and activity modules and attend online LC group sessions over 90 minutes once weekly (QW) for 8 weeks. Patients receive informational emails weekly prior to scheduled sessions.

GROUP 3 (ACLP-LC-IHC): Patients participate in the 8-week ACLP-LC program just like group 2. In addition, starting two weeks after the end of the program, they receive IHC sessions over 30-60 minutes for up to 6 sessions over 3 months.

Additionally, patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HR+/HER2 negative MBC
2. On first- or second-line treatment
3. Life expectancy at least 12 months
4. Only females
5. Age 18 years or older
6. Able to read, write, and speak English
7. Willingness to follow protocol requirements
8. Have a smartphone with access to cellular service or computer access with internet service
9. Oriented to person, place, and time
10. Consume less than 3 servings of fruit and vegetable/day
11. Engage in less than 150 minutes moderate/vigorous intensity activity per week, defined as anything that causes small increases in breathing or heart rate for a sustained amount of time (e.g., brisk walking, bicycling)
12. Engage in a mind-body practice less than 4 times a month

Exclusion Criteria:

1. Another primary cancer diagnosis within past 5 years (not including non-melanoma skin cancers)
2. Any major thought disorder (e.g., schizophrenia, dementia)
3. Communication barriers (e.g., hard of hearing)
4. Poorly-controlled or uncontrolled diabetes in the opinion of the physician(s)
5. Extreme mobility issues (e.g., unable to get in and out of a chair unassisted)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Meroe Morse, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org